CLINICAL TRIAL: NCT04545099
Title: Comparison of the Impacts of Sugammadex With Neostigmine on Patency of Laryngeal Opening (Glottic Aperture Angle)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4-2020-0804
Record Dates: First submitted 2020-09-01; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Supraglottic Airway Device Insertion
MeSH Terms: interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: triple (Participant, Care Provider, investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sugammadex (Experimental): Administration of Sugammadex
  Interventions: Drug: Sugammadex
- Neostigmine (Active Comparator): Administration of Neostigmine
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Sugammadex — Administration of Sugammadex for muscle relaxation reversal
  Arms: Sugammadex
Drug: Neostigmine — Administration of Neostigmine for muscle relaxation reversal
  Arms: Neostigmine

SUMMARY:
The aim of this study is to compare the degree of change in the angle of the vocal cords before and after administration of neostigmine or sugammadex. Moreover, we intend to compare the angle of vocal folds after administration of neostigmine or sugammadex.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients who undergoes elective surgery under general anesthesia with supraglottic airway device.

Exclusion Criteria:

1. Patients under 20 years old
2. Pregnant women
3. Patients who can not read the consent form or are not fluent in Korean (illiterate, foreigner)
4. Patients who refused the clinical trial
5. Patients with dementia or cognitive impairment
6. Patients with neuromuscular disorders impairing neuromuscular blockade
7. Renal dysfunction (estimated Glomerular Filtration Rate less than 30 ml/min/1.73m2)
8. Past history of allergic reactions to neostigmine or sugammadex
9. Patients with ASA class IV or higher
10. Robotic surgery, adenoid or tonsillectomy
11. Patients with moderate or severe asthma, pulmonary function tests with forced expiratory volume for 1second of 1 liter or less, patients with upper respiratory infection symptoms within 2 weeks before surgery, current smokers (within 1 month of smoking cessation is included.)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Angle of vocal folds after administration of sugammadex or neostigmine 2) Degree of change in angle of vocal folds before and after administration of sugammadex or neostigmine | 1-2 minutes after drug administration (inhalation, exhalation)
Degree of change in angle of vocal folds before and after administration of sugammadex or neostigmine | 1) Just before drug administration 2) 1-2 minutes after drug administration (inhalation, exhalation)

SECONDARY OUTCOMES:
Time to recover from spontaneous breathing | immediately after drug(sugammadex or neostigmine) administration
  Time taken to recover from spontaneous breathing(6ml/kg or more) after administration of sugammadex or neostigmine
Time to extubation | immediately after drug(sugammadex or neostigmine) administration
  Time taken to extubation after administration of sugammadex or neostigmine

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Rim Lee, Principal Investigator — Severance Hospital

IPD SHARING:
Plan to Share IPD: Undecided